CLINICAL TRIAL: NCT02080520
Title: Nattokinase Atherothrombotic Prevention Study
Acronym: NAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Howard N. Hodis, M.D., Harry J Bauer and Dorothy Bauer Rawlins Professor of Cardiology, Professor of Medicine, Population and Public Health Sciences, and Molecular Pharmacology and Toxicology, Director, Atherosclerosis Research Unit, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SDF-01
Record Dates: First submitted 2014-02-21; First posted 2014-03-06 (Estimated); Results first posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Prevention of Subclinical Atherosclerosis Progression; Prevention of Cognitive Decline
Keywords: Arterial compliance; Arterial distensibility; Atherosclerosis; Atherothrombosis; Blood pressure; Cardiovascular disease (CVD); Carotid artery; Carotid artery intima-media thickness (CIMT); Coagulation; Cognition; Fermented soy; Fibrinolysis; Natto; Nattokinase; Prevention; Randomized controlled trial; Rheology; Soy; Soybeans; Thrombosis
MeSH Terms: conditions — Atherosclerosis; Thrombosis; Cardiovascular Diseases | interventions — nattokinase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nattokinase (Active Comparator): Oral nattokinase 2,000 fibrinolytic units daily
  Interventions: Dietary Supplement: Nattokinase
- Placebo (Placebo Comparator): Matched placebo daily
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Nattokinase
  Arms: Nattokinase
Other: Placebo
  Arms: Placebo

SUMMARY:
The potential for nattokinase to "thin" blood and to reduce blood clotting by positive antithrombotic and fibrinolytic effects presents a unique opportunity to safely study such effects on cardiovascular disease and cognition. Unfortunately, such studies of antithrombotic and fibrinolytic pathways of prevention have been limited due to lack of safe compounds and the adverse reactions associated with current agents such as Coumadin. Nattokinase, an over-the-counter supplement used for cardiovascular health, is the most active functional constituent of natto, a fermented soy product. Natto has been consumed primarily by the Japanese for over 1000 years, a population with one of the lowest risks for cardiovascular disease and dementia. Cardiovascular disease and dementia remain the most challenging age-related health risks of the 21st century for Americans necessitating development of further effective preemptive strategies. Whether reducing the propensity for thrombus formation and/or increasing fibrinolytic activity can prevent the progression of atherosclerosis and cognitive decline has not yet been determined.

Using nattokinase under primary prevention conditions, the investigators propose to conduct a randomized, double-blinded, placebo-controlled trial to determine whether decreasing atherothrombotic risk can reduce the progression of subclinical atherosclerosis and cognitive decline. The investigators propose to randomize 240 healthy non-demented women and men to nattokinase supplementation or to placebo for three years. The primary trial endpoints will be measurement of carotid arterial wall thickness and arterial stiffness, early changes of atherosclerosis that can be measured safely by non-invasive imaging techniques. The secondary trial endpoint will be ascertained through change in cognition measured by a neuropsychological battery. In addition, biochemical blood measurements and in vitro studies will be conducted to compare the effects of nattokinase relative to placebo on blood coagulation and thrombus break-down capabilities, blood flow properties, inflammation and inflammatory activation of endothelial cells that line blood vessels.

DETAILED DESCRIPTION:
Objectives and Hypotheses: The goal of the proposed study is to determine under randomized controlled trial (RCT) conditions whether nattokinase supplementation reduces subclinical atherosclerosis progression and cognitive decline in healthy women and men. The investigators' hypotheses are: 1) Compared to placebo, nattokinase supplementation will show less subclinical atherosclerosis progression and cognitive decline in healthy women and men; 2) The reduction in subclinical atherosclerosis progression and cognitive decline with nattokinase supplementation will be correlated; and, 3) The reduction in progression of subclinical atherosclerosis and cognitive decline with nattokinase supplementation will be mediated through hemostatic, fibrinolytic, and hemorheological factors as well as attenuation of inflammation, monocyte activation, vascular endothelium injury, and activation of vascular endothelium by circulating monocytes.

Specific Aims: To conduct a RCT to determine the effect of nattokinase supplementation on the progression of subclinical atherosclerosis (primary trial end point) and cognitive decline (secondary trial end point). Healthy non-demented women and men >55 years old without pre-existing symptomatic CVD and diabetes mellitus will be randomized over a 2-year period to oral nattokinase (2,000 fibrinolysis units) daily versus placebo in this double-blind, placebo-controlled trial; randomized treatment will be 3-years. The following 5 major specific aims will be completed:

To determine the effect of nattokinase supplementation on progression of subclinical carotid artery atherosclerosis determined as the rate of change of the common carotid artery intima-media thickness (CIMT) and arterial stiffness in computer image processed B-mode ultrasonograms.

To determine the effect of nattokinase supplementation on cognitive decline determined with a neuropsychological battery designed to evaluate 7 cognitive domains including: attention, concentration, working memory, executive function; visuospatial/visuoconstructive skills; naming/semantic memory; and verbal and nonverbal episodic memory.

To determine the effect of nattokinase supplementation on cognitive decline according to apolipoprotein (Apo) E4 genotype.

To determine the association of subclinical atherosclerosis progression with cognitive decline.

To determine whether the effects of nattokinase supplementation on subclinical atherosclerosis and cognitive decline are mediated through hemostatic (fibrinogen, factor VIII, platelet activity), fibrinolytic (tPA, PAI-1, D-dimer), hemorheological (plasma and blood viscosity, red blood cell aggregation), and inflammatory (MCP-1, IL-8, TNFα, IL-1β, IL-10, monocyte cell surface markers CD11b/CD11c and VLA-4, and cellular adhesion molecules VCAM-1 and ICAM-1) factors as well as blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Age >55 years
* Male or postmenopausal female (no uterine bleeding for >6 months)

Exclusion Criteria:

* Clinical signs, symptoms, or personal history of cardiovascular disease
* Diabetes mellitus or fasting serum glucose >140 mg/dL
* Plasma triglyceride levels >500 mg/dL
* Uncontrolled hypertension (systolic blood pressure >160 mmHg or diastolic blood pressure >110 mmHg)
* Uncontrolled tachycardia or irregular heart rates (i.e., atrial fibrillation)
* Thyroid disease (untreated)
* Renal insufficiency (defined as serum creatinine >2.0 mg/dL)
* Life threatening illness with prognosis <5 years
* Current use of lipid-lowering medication
* Current use of food supplements containing soy, soy protein, isoflavones or other phytoestrogens
* Known sensitivity or allergy to soy or nuts
* Regular aspirin or other antiplatelet medication use
* Use of anticoagulants
* Bleeding diatheses or tendencies

Ages: 55 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2014-04; Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard N. Hodis, M.D., Principal Investigator — Atherosclerosis Research Unit, University of Southern California
Locations (1):
- Atherosclerosis Research Unit, University of Southern California, Los Angeles, California, United States

REFERENCES:
- [Result] Hodis HN, Mack WJ, Meiselman HJ, Kalra V, Liebman H, Hwang-Levine J, Dustin L, Kono N, Mert M, Wenby RB, Huesca E, Rochanda L, Li Y, Yan M, St John JA, Whitfield L. Nattokinase atherothrombotic prevention study: A randomized controlled trial. Clin Hemorheol Microcirc. 2021;78(4):339-353. doi: 10.3233/CH-211147. PMID 33843667

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the general population through media campaigns.
Pre-assignment Details: 1189 individuals were screened by telephone, 857 did not meet inclusion criteria. 332 individuals were screened in research clinic, 67 were excluded (51 did not meet inclusion criteria; 16 declined to participate). 265 individuals were randomized.
Groups:
- Placebo: Matching placebo daily
Period: Overall Study
Arm/Group | Nattokinase | Placebo
Started | 132 | 133
Completed | 118 | 116
Not Completed | 14 | 17
Not completed — Self-reported symptoms | 5 | 6
Not completed — Unable to contact | 2 | 1
Not completed — Initiated aspirin | 2 | 0
Not completed — Atrial fibrillation | 1 | 1
Not completed — Cancer | 1 | 2
Not completed — Not interested in study | 1 | 3
Not completed — Too busy | 1 | 1
Not completed — Work-related injury | 1 | 0
Not completed — Personal reasons | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nattokinase | Placebo | Total
Number analyzed (Participants) | 132 | 133 | 265
Age, Customized [Median (Inter-Quartile Range); unit: years] | 65.4 [60.8 to 72.3] | 65.2 [60.6 to 71.7] | 65.3 [60.7 to 71.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 81 | 164
  Male | 49 | 52 | 101
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, non-Hispanic | 94 | 93 | 187
  Black, non-Hispanic | 11 | 4 | 15
  Asian, non-Hispanic | 10 | 15 | 25
  Hispanic | 16 | 19 | 35
  Other | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 132 | 133 | 265

OUTCOME MEASURES:

1. Primary Outcome: Progression of Subclinical Atherosclerosis
Description: Rate of change in distal common carotid artery (CCA) far wall intima-media thickness (mm per year) in computer image processed B-mode ultrasonograms will be a co-primary trial endpoint.
Time Frame: Baseline x 2 and then every 6 months, up to 3 years
Measure: Mean (95% Confidence Interval); unit: mm per year
Arm/Group | Nattokinase | Placebo
Number analyzed (Participants) | 132 | 133
mm per year | 0.013 [0.010 to 0.015] | 0.011 [0.009 to 0.013]
Statistical Analysis 1: Comparison: Nattokinase vs Placebo; Test type: Superiority; p = 0.31, Mixed Models Analysis

2. Primary Outcome: Progression of Carotid Artery Stiffness (Distensibility)
Description: Rate of change in arterial distensibility of the distal common carotid artery (CCA) determined from lumen diameters at systole and diastole and systolic and diastolic blood pressure. CCA lumen diameters will be determined from computer image processed B-mode ultrasonograms. This is a co-primary trial endpoint.
Time Frame: Baseline x 2 and then every 6 months, up to 3 years
Measure: Mean (95% Confidence Interval); unit: x(10^-6)(N^-1)(m^2) per year
Arm/Group | Nattokinase | Placebo
Number analyzed (Participants) | 132 | 133
x(10^-6)(N^-1)(m^2) per year | -0.501 [-0.742 to -0.261] | -0.389 [-0.633 to -0.144]
Statistical Analysis 1: Comparison: Nattokinase vs Placebo; Test type: Superiority; p = 0.52, Mixed Models Analysis

3. Primary Outcome: Carotid Artery Stiffness Progression (Compliance)
Description: Rate of change in arterial compliance of the distal common carotid artery (CCA) determined from lumen diameters at systole and diastole and systolic and diastolic blood pressure. CCA lumen diameters will be determined from computer image processed B-mode ultrasonograms. This is a co-primary trial endpoint.
Time Frame: Baseline x 2 and then every 6 months, up to 3 years
Measure: Mean (95% Confidence Interval); unit: mm^2/kPa per year
Arm/Group | Nattokinase | Placebo
Number analyzed (Participants) | 132 | 133
mm^2/kPa per year | -0.019 [-0.032 to -0.007] | -0.010 [-0.023 to 0.002]
Statistical Analysis 1: Comparison: Nattokinase vs Placebo; Test type: Superiority; p = 0.32, Mixed Models Analysis

4. Secondary Outcome: Change in Neurocognitive Function (Global Cognition)
Description: All neuropsychological test scores at baseline and follow-up assessments were standardized ([raw score - mean score]/standard deviation) using the baseline means and standard deviations from the entire NAPS sample. Each of three cognitive composite scores was calculated at baseline (composite score of 0 equals performance at the mean of each test at baseline) and follow-up assessments as the weighted average of the individual donor standardized test scores, weighted by the inverse correlation among tests. The change from baseline (endpoint minus baseline cognitive outcome) was computed for each of the cognitive composite scores (verbal memory, global cognition, and executive functions). Since the outcome is not a single test but a weighted average of multiple tests, the range is not standard and not reported and there is no clinically relevant threshold. A composite score and change in composite score greater than 0 represent better cognitive performance.
Time Frame: Baseline and 36 months
Measure: Mean (95% Confidence Interval); unit: Z-score
Groups:
- Nattokinase: Oral nattokinase 2,000 fibrinolytic units daily
  Nattokinase
- Placebo: Matched placebo daily
  Placebo
Arm/Group | Nattokinase | Placebo
Number analyzed (Participants) | 132 | 133
Z-score | 0.43 [0.22 to 0.63] | 0.43 [0.22 to 0.64]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for up to 3 years for each participant.
Arm/Group | Nattokinase | Placebo
All-Cause Mortality (participants affected / at risk) | 0/132 | 1/133
Serious Adverse Events (participants affected / at risk) | 13/132 | 15/133
Other Adverse Events (participants affected / at risk) | 58/132 | 57/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nattokinase (N=132) | Placebo (N=133)
Pancreatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Non-fatal myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Chest pain (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery bypass graft surgery (Surgical and medical procedures) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Transient ischemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Breast ductal carcinoma in-situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast invasive ductal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Follicular lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 1 (1) | 2 (2)
Radical prostatectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hip fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Perforated appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Carotid endarterectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Benign tumor excision (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nattokinase (N=132) | Placebo (N=133)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thymic cyst (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 2 (2)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 2 (2)
Cataract (Eye disorders) | 1 (2) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 3 (3)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colon polyps (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 2 (2)
Multiple allergies (Immune system disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (3)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Dermatitis contact (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Angiogram (Investigations) | 1 (1) | 1 (1)
Arteriogram coronary (Investigations) | 0 (0) | 1 (1)
Arthroscopy (Investigations) | 1 (1) | 1 (1)
Biopsy (Investigations) | 1 (1) | 0 (0)
Biopsy breast (Investigations) | 0 (0) | 2 (2)
Biopsy colon (Investigations) | 1 (2) | 0 (0)
Biopsy prostate (Investigations) | 1 (1) | 0 (0)
Biopsy skin (Investigations) | 1 (1) | 0 (0)
Biopsy thyroid gland (Investigations) | 0 (0) | 1 (1)
Colonoscopy (Investigations) | 3 (3) | 0 (0)
Weight increased (Investigations) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (6) | 4 (4)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Osteochondroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 2 (2) | 0 (0)
Dementia Alzheimer's type (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 2 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Parkinson's disease (Nervous system disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Libido decreased (Psychiatric disorders) | 1 (1) | 0 (0)
Ureterolithiasis and Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Breast cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast tenderness (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Hot flush (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Apicoectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Appendicectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Breast prosthesis implantation (Surgical and medical procedures) | 0 (0) | 1 (1)
Bunion and toe operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Bunion operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Cardiac ablation (Surgical and medical procedures) | 0 (0) | 1 (1)
Cardiac pacemaker insertion (Surgical and medical procedures) | 1 (1) | 1 (1)
Cataract operation (Surgical and medical procedures) | 3 (4) | 1 (1)
Dental implantation (Surgical and medical procedures) | 0 (0) | 1 (1)
Dupuytren's contracture operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Eyelid operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Femoral hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Haemorrhoid operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 1 (1) | 1 (1)
Inguinal hernia repair (Surgical and medical procedures) | 1 (1) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 2 (2) | 2 (2)
Knee operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Large intestinal polypectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Meniscus operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Oesophagogastric fundoplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Prostatic radiotherapies (Surgical and medical procedures) | 0 (0) | 1 (1)
Rotator cuff repair (Surgical and medical procedures) | 2 (2) | 0 (0)
Shoulder arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Spinal laminectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgery, hernia (Surgical and medical procedures) | 1 (1) | 0 (0)
Suture insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Tendon sheath incision (Surgical and medical procedures) | 1 (1) | 0 (0)
Thyroidectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Trapeziectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Vitrectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-03-10): https://cdn.clinicaltrials.gov/large-docs/20/NCT02080520/Prot_SAP_000.pdf